CLINICAL TRIAL: NCT00432666
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Multi-center Trial With an Open-label Extension Period to Investigate the Efficacy and Safety of incobotulinumtoxinA (Xeomin) in the Treatment of Post-stroke Spasticity of the Upper Limb
Brief Title: IncobotulinumtoxinA (Xeomin) Versus Placebo in the Treatment of Post-stroke Spasticity of the Upper Limb
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Clinical R&D CNS, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ 60201-0410
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Post-stroke Upper Limb Spasticity
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IncobotulinumtoxinA (Xeomin) (Experimental): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), up to five injections in the Open-Label Extension Period, up to 400 units at each injection visit; Mode of administration: intramuscular injection
  Interventions: Drug: IncobotulinumtoxinA (Xeomin)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin) — incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), up to five injections in the Open-Label Extension Period, up to 400 units at each injection visit; Mode of administration: intramuscular injection
  Arms: IncobotulinumtoxinA (Xeomin)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
IncobotulinumtoxinA (Xeomin) is a botulinum toxin type A preparation free from complexing proteins, i.e. free from proteins other than the active toxin. Injected into the muscle, incobotulinumtoxinA (Xeomin) causes local weakening. Botulinum toxin type A is widely used for treatment of various neurological conditions. This study will investigate the efficacy and safety of incobotulinumtoxinA (Xeomin) in the treatment of post-stroke spasticity of the upper limb.

ELIGIBILITY:
Main Inclusion Criteria:

* Female or male patients ≥ 18 years
* ≥ 6 months since the last stroke, diagnosed by an appropriate health care professional (e.g., neurologist)
* Focal spasticity with ≥ 2 points on the Ashworth Scale in the wrist flexors with clinical pattern Flexed Wrist
* Focal spasticity with ≥ 2 points on the Ashworth Scale in the fingers flexors with clinical pattern Clenched Fist
* For pre-treated patients only: source documentation of the most recent injection session with Botulinum Toxin and sufficient therapeutic response for Flexed Wrist and Clenched Fist
* For pre-treated patients only: the most recent injection with Botulinum Toxin must have been maximal 50 Units BOTOX® or 200 Units Dysport® or 2000 Units Neurobloc® (type B preparation) per each of these flexors: carpi ulnaris, digitorum superficialis, digitorum profundus
* For pre-treated patients only: the most recent injection with Botulinum Toxin must have been maximal 60 Units BOTOX® or 240 Units Dysport® or 2400 Units Neurobloc® (type B preparation) for flexor carpi radialis

Main Exclusion Criteria:

* Spasticity of any other origin than stroke
* Previous treatment with Botulinum Toxin of any serotype and for any body region within the 4 months prior to Screening (Visit 1, Day -7)
* Planned concomitant treatment with Botulinum Toxin of any serotype and for any body region
* Previous or planned treatment with phenol- or alcohol-injection in the target limb
* Previous surgical treatment of spasticity in the target muscle(s)
* Fixed contracture, defined as severe restriction of the range of joint movement on passive stretch
* Severe atrophy of the target limb muscles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2006-06; Primary Completion 2006-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Pharmaceuticals, Study Chair — Merz Pharmaceuticals GmbH
Locations (3):
- Czech Republic, Czechia
- Hungary, Hungary
- Poland, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- incobotulinumtoxinA (Xeomin): incobotulinumtoxinA (Xeomin) (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection
- Placebo: Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection Dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl; Mode of administration: intramuscular injection
Period: Main Period
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Started | 73 | 75
Completed | 71 | 74
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Consent Withdrawn | 1 | 0
Period: Open-Label Extension Period
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Started | 145 | 0 (In the Open-Label Extension Period no placebo treatment arm was given.)
Completed | 120 | 0
Not Completed | 25 | 0
Not completed — Withdrawal Criteria Occurred | 1 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Consent withdrawn | 10 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo | Total
Number analyzed (Participants) | 73 | 75 | 148
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.2) | 53.3 (13.3) | 55.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 45 | 50 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction of at Least 1 Point at Week 4 Compared to Baseline in Ashworth Score in Wrist Flexors
Description: The Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension). Subjects with a reduction of one point were defined as responder for the aim of the primary efficacy analysis.
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects; missing values were not imputed
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants | 50 | 28
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) vs Placebo; The null hypothesis was equality of the chance (OR = 1) for a clinically relevant treatment effect between incobotulinumtoxinA (Xeomin) and placebo at Week 4 for wrist flexors. Responders were defined as subjects with an improvement of at least 1 point in the Ashworth score compared with Baseline. The dependent variable was the response to treatment, the independent variables were treatment, Ashworth score at the Baseline Visit, pre-treated patient status, gender, age, BMI, and pooled sites; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.97, 95% CI 2-sided [1.90 to 8.30], Standard Error of Mean 1.49

2. Secondary Outcome: Responders at Week 4 Based on a Responder Definition of at Least 2 Points Improvement From Baseline in the Ashworth Score for Wrist Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects; missing values were imputed by worst case, i.e. zero change
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants | 14 | 3

3. Secondary Outcome: Responders Based on a Responder Definition of at Least 1 Point Improvement From Baseline in the Ashworth Score for Wrist Flexors at All Other Post Baseline Visits
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 8, Week 12, Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Week 2 | 45 | 22
  Week 8 | 49 | 22
  Week 12 | 31 | 18
  Final Visit | 29 | 14

4. Secondary Outcome: Responders Based on a Responder Definition of at Least 1 Point Improvement From Baseline in the Ashworth Score for Treated Elbow Flexors at All Post Baseline Visits
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Week 2 | 32 | 15
  Week 4 | 34 | 21
  Week 8 | 27 | 22
  Week 12 | 23 | 16
  Final Visit | 21 | 14

5. Secondary Outcome: Responders Based on a Responder Definition of at Least 1 Point Improvement From Baseline in the Ashworth Score for Treated Forearm Pronators at All Post Baseline Visits
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Week 2 | 16 | 10
  Week 4 | 19 | 12
  Week 8 | 18 | 11
  Week 12 | 12 | 11
  Final Visit | 10 | 9

6. Secondary Outcome: Responders Based on a Responder Definition of at Least 1 Point Improvement From Baseline in the Ashworth Score for Treated Finger Flexors at All Post Baseline Visits
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Week 2 | 50 | 22
  Week 4 | 50 | 27
  Week 8 | 44 | 27
  Week 12 | 35 | 23
  Final Visit | 28 | 17

7. Secondary Outcome: Responders Based on a Responder Definition of at Least 1 Point Improvement From Baseline in the Ashworth Score for Treated Thumb Flexors at All Post Baseline Visits
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Week 2 | 16 | 8
  Week 4 | 17 | 11
  Week 8 | 14 | 14
  Week 12 | 14 | 10
  Final Visit | 11 | 10

8. Secondary Outcome: Change From Baseline to Week 2 in Ashworth Scale Score for Treated Elbow Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 5 | 0
  Change of "-1" points | 27 | 15
  Change of "0" points | 22 | 39
  Change of "+1" points | 0 | 1

9. Secondary Outcome: Change From Baseline to Week 4 in Ashworth Scale Score for Treated Elbow Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 5 | 1
  Change of "-1" points | 29 | 20
  Change of "0" points | 20 | 32
  Change of "+1" points | 0 | 2

10. Secondary Outcome: Change From Baseline to Week 8 in Ashworth Scale Score for Treated Elbow Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 6 | 2
  Change of "-1" points | 20 | 20
  Change of "0" points | 26 | 31
  Change of "+1" points | 0 | 2
  Missing | 1 | 0

11. Secondary Outcome: Change From Baseline to Week 12 in Ashworth Scale Score for Treated Elbow Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 5 | 0
  Change of "-1" points | 18 | 16
  Change of "0" points | 31 | 36
  Change of "+1" points | 0 | 2
  Missing | 0 | 1

12. Secondary Outcome: Change From Baseline to Final Visit in Ashworth Scale Score for Treated Elbow Flexors
Description: as for outcome 1
Time Frame: Baseline, Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 54 | 55
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 19 | 14
  Change of "0" points | 32 | 37
  Change of "+1" points | 1 | 3
  Missing | 0 | 1

13. Secondary Outcome: Change From Baseline to Week 2 in Ashworth Scale Score for Treated Forearm Pronators
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 3 | 0
  Change of "-1" points | 13 | 10
  Change of "0" points | 18 | 27
  Change of "+1" points | 1 | 1

14. Secondary Outcome: Change From Baseline to Week 4 in Ashworth Scale Score for Treated Forearm Pronators
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 16 | 12
  Change of "0" points | 16 | 24
  Change of "+1" points | 0 | 1
  Missing | 0 | 1

15. Secondary Outcome: Change From Baseline to Week 8 in Ashworth Scale Score for Treated Forearm Pronators
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 15 | 11
  Change of "0" points | 16 | 25
  Change of "+1" points | 1 | 1
  Missing | 0 | 1

16. Secondary Outcome: Change From Baseline to Week 12 in Ashworth Scale Score for Treated Forearm Pronators
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 10 | 11
  Change of "0" points | 21 | 20
  Change of "+1" points | 1 | 5
  Missing | 1 | 2

17. Secondary Outcome: Change From Baseline to Final Visit in Ashworth Scale Score for Treated Forearm Pronators
Description: as for outcome 1
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 35 | 38
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 1 | 1
  Change of "-1" points | 9 | 8
  Change of "0" points | 22 | 21
  Change of "+1" points | 2 | 6
  Missing | 1 | 2

18. Secondary Outcome: Change From Baseline to Week 2 in Ashworth Scale Score for Wrist Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 11 | 2
  Change of "-1" points | 33 | 20
  Change of "0" points | 27 | 51
  Change of "+1" points | 1 | 0

19. Secondary Outcome: Change From Baseline to Week 4 in Ashworth Scale Score for Wrist Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 13 | 3
  Change of "-1" points | 36 | 25
  Change of "0" points | 22 | 41
  Change of "+1" points | 1 | 3
  Missing | 0 | 1

20. Secondary Outcome: Change From Baseline to Week 8 in Ashworth Scale Score for Wrist Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 13 | 4
  Change of "-1" points | 35 | 18
  Change of "0" points | 21 | 47
  Change of "+1" points | 2 | 3
  Missing | 1 | 1

21. Secondary Outcome: Change From Baseline to Week 12 in Ashworth Scale Score for Wrist Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 9 | 2
  Change of "-1" points | 21 | 16
  Change of "0" points | 38 | 47
  Change of "+1" points | 2 | 6
  Missing | 2 | 2

22. Secondary Outcome: Change From Baseline to Final Visit in Ashworth Scale Score for Wrist Flexors
Description: as for outcome 1
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 73
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 27 | 14
  Change of "0" points | 39 | 50
  Change of "+1" points | 4 | 7
  Missing | 1 | 2

23. Secondary Outcome: Change From Baseline to Week 2 in Ashworth Scale Score for Finger Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 4 | 0
  Change of "-2" points | 8 | 2
  Change of "-1" points | 38 | 20
  Change of "0" points | 21 | 50
  Change of "+1" points | 2 | 3

24. Secondary Outcome: Change From Baseline to Week 4 in Ashworth Scale Score for Finger Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 5 | 0
  Change of "-2" points | 15 | 5
  Change of "-1" points | 30 | 22
  Change of "0" points | 22 | 44
  Change of "+1" points | 1 | 3
  Missing | 0 | 1

25. Secondary Outcome: Change From Baseline to Week 8 in Ashworth Scale Score for Finger Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 18 | 3
  Change of "-1" points | 24 | 24
  Change of "0" points | 27 | 43
  Change of "+1" points | 1 | 4
  Missing | 1 | 1

26. Secondary Outcome: Change From Baseline to Week 12 in Ashworth Scale Score for Finger Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 9 | 2
  Change of "-1" points | 24 | 21
  Change of "0" points | 33 | 45
  Change of "+1" points | 3 | 5
  Missing | 2 | 2

27. Secondary Outcome: Change From Baseline to Final Visit in Ashworth Scale Score for Finger Flexors
Description: as for outcome 1
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 1
  Change of "-1" points | 26 | 16
  Change of "0" points | 39 | 51
  Change of "+1" points | 5 | 5
  Missing | 1 | 2

28. Secondary Outcome: Change From Baseline to Week 2 in Ashworth Scale Score for Treated Thumb Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 3 | 1
  Change of "-1" points | 13 | 7
  Change of "0" points | 10 | 22
  Change of "+1" points | 0 | 1

29. Secondary Outcome: Change From Baseline to Week 4 in Ashworth Scale Score for Treated Thumb Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 6 | 2
  Change of "-1" points | 11 | 9
  Change of "0" points | 9 | 18
  Change of "+1" points | 0 | 1
  Missing | 0 | 1

30. Secondary Outcome: Change From Baseline to Week 8 in Ashworth Scale Score for Treated Thumb Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 6 | 2
  Change of "-1" points | 8 | 12
  Change of "0" points | 11 | 15
  Change of "+1" points | 1 | 0
  Change of "+2" points | 0 | 1
  Missing | 0 | 1

31. Secondary Outcome: Change From Baseline to Week 12 in Ashworth Scale Score for Treated Thumb Flexors
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Change of "-3" points | 0 | 1
  Change of "-2" points | 4 | 1
  Change of "-1" points | 10 | 8
  Change of "0" points | 11 | 14
  Change of "+1" points | 0 | 4
  Change of "+2" points | 0 | 1
  Missing | 1 | 2

32. Secondary Outcome: Change From Baseline to Final Visit in Ashworth Scale Score for Treated Thumb Flexors
Description: as for outcome 1
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Change of "-3" points | 0 | 1
  Change of "-2" points | 2 | 0
  Change of "-1" points | 9 | 9
  Change of "0" points | 13 | 14
  Change of "+1" points | 1 | 4
  Change of "+2" points | 0 | 1
  Missing | 1 | 2

33. Secondary Outcome: Time to Onset of Treatment Effect
Description: Starting with the visit 2 weeks after baseline injection the subject was asked if he/she experienced an treatment effect and if "yes": when. If the subject did not experience an treatment effect he/she was asked again at each of the following visits (at week 4, 8, and 12) of the Main Period until the answer was "yes" or until the final visit of the Main Period was performed.
  For subjects without any treatment effect the time to onset of effect was censored at the last visit of the Main Period.
Time Frame: Period starting at Visit 2 (baseline injection) of the Main Period up to onset of treatment effect
Population: Results for placebo patients were not displayed because the upper limit of the confidence interval was not estimable (this can not be entered because a numeric entry is expected). The results of this analysis are therefore given as "Onset of Treatment Effect [classified]" under "Other Pre-specified Outcome".
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 0
Days | 4.0 [3.0 to 7.0] |

34. Secondary Outcome: Time to Waning of Treatment Effect
Description: Subject who reported an onset of treatment effect were asked at each visit/telephone contact starting at week 4 at earliest if he/she felt that there was a waning of the treatment effect. The same question was asked at each of the following telephone contacts and visits (up to the Final Visit of the Main Period) if the answer at the respective previous visit was "no". If the patient answered with "yes" he/she will be asked at which week after the injection (= the time span in weeks) the waning of effect occurred. For all subjects without an onset of treatment effect the waning was set to zero.
Time Frame: Defined as time (weeks) from Visit 2 (injection session at Baseline, Day 0) to the subjective estimation of the waning of the effect
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Weeks | 10.0 [9.0 to 11.0] | 10.0 [10.0 to 11.0]

35. Secondary Outcome: Duration of Treatment Effect
Description: The duration of treatment effect is defined as the time period from the day of injection until the time point of a need for a new injection agreed by the patient and the investigator. For subjects without any treatment effect the duration of effect was set to zero.
Time Frame: Period from the day of injection until the time point of a need for a new injection agreed by the patient and the investigator
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Days | 87.0 [86.0 to 94.0] | 84.0 [0.0 to 84.0]

36. Other Pre Specified Outcome: Onset of Treatment Effect [Classified]
Description: as for outcome 33
Time Frame: Period starting at baseline injection of the Main Period up to onset of treatment effect
Population: These results are a different presentation of the results of the secondary outcome measure "Time to Onset of Treatment Effect". For subjects without any treatment effect the time to onset of effect was censored at the last visit.
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Onset at Day 1, 2 or 3 | 32 | 14
  Onset at Day 4, 5 or 6 | 12 | 4
  Onset at Day 7, 8 or 9 | 9 | 11
  Onset at Day 10, 11 or 12 | 1 | 6
  Onset at Day 13, 14 or 15 | 3 | 1
  Onset at Day 16, 17 or 18 | 1 | 1
  Onset at Day 19, 20 or 21 | 3 | 3
  Onset at Day 22, 23 or 24 | 0 | 2
  Onset later than Day 25 | 2 | 1
  Censored | 10 | 32

37. Secondary Outcome: Investigator's Global Assessment of Efficacy
Description: The Investigator's Global Assessment of Efficacy is a subjective estimation assessed on a 4-point Likert scale with the items 1=very good, 2=good, 3=moderate, and 4=poor.
Time Frame: Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Very good | 11 | 2
  Good | 32 | 24
  Moderate | 14 | 12
  Poor | 15 | 35
  Missing | 1 | 2

38. Secondary Outcome: Patient's Global Assessment of Efficacy
Description: The Patient's Global Assessment of Efficacy is a subjective estimation assessed on a 4-point Likert scale with the items 1=very good, 2=good, 3=moderate, and 4=poor.
Time Frame: Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Very good | 7 | 2
  Good | 41 | 21
  Moderate | 9 | 17
  Poor | 15 | 33
  Missing | 1 | 2

39. Secondary Outcome: Carer's Global Assessment of Efficacy
Description: The Carer's Global Assessment of Efficacy is a subjective estimation assessed on a 4-point Likert scale with the items 1=very good, 2=good, 3=moderate, and 4=poor.
Time Frame: Final Visit of the Main Period (to be performed at week 12 after 1st injection at earliest, at week 20 at latest)
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Very good | 8 | 2
  Good | 21 | 17
  Moderate | 9 | 10
  Poor | 8 | 24
  No carer | 26 | 19
  Missing | 1 | 3

40. Secondary Outcome: Change From Baseline to Week 2 in the Disability Assessment Scale for the Principal Therapeutic Target
Description: The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 7 | 1
  Change of "-1" points | 21 | 8
  Change of "0" points | 43 | 66
  Change of "+1" points | 2 | 0
  Change of "+2" points | 0 | 0

41. Secondary Outcome: Change From Baseline to Week 4 in the Disability Assessment Scale for the Principal Therapeutic Target
Description: as for outcome 40
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 12 | 1
  Change of "-1" points | 21 | 15
  Change of "0" points | 40 | 57
  Change of "+1" points | 1 | 1
  Change of "+2" points | 0 | 0
  Missing | 0 | 1

42. Secondary Outcome: Change From Baseline to Week 8 in the Disability Assessment Scale for the Principal Therapeutic Target
Description: as for outcome 40
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 6 | 1
  Change of "-1" points | 26 | 15
  Change of "0" points | 37 | 57
  Change of "+1" points | 2 | 1
  Change of "+2" points | 0 | 0
  Missing | 2 | 1

43. Secondary Outcome: Change From Baseline to Week 12 in the Disability Assessment Scale for the Principal Therapeutic Target
Description: as for outcome 40
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 3 | 2
  Change of "-1" points | 24 | 10
  Change of "0" points | 42 | 58
  Change of "+1" points | 2 | 3
  Change of "+2" points | 0 | 0
  Missing | 2 | 2

44. Secondary Outcome: Change From Baseline to Final Visit in the Disability Assessment Scale for the Principal Therapeutic Target
Description: as for outcome 40
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 1
  Change of "-1" points | 20 | 14
  Change of "0" points | 47 | 55
  Change of "+1" points | 2 | 3
  Change of "+2" points | 1 | 0
  Missing | 2 | 2

45. Secondary Outcome: Change From Baseline to Week 2 in the Disability Assessment Scale for Domain "Hygiene"
Description: as for outcome 40
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 6 | 1
  Change of "-1" points | 12 | 7
  Change of "0" points | 52 | 66
  Change of "+1" points | 1 | 1
  Change of "+2" points | 0 | 0

46. Secondary Outcome: Change From Baseline to Week 4 in the Disability Assessment Scale for Domain "Hygiene"
Description: as for outcome 40
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 3 | 0
  Change of "-2" points | 5 | 1
  Change of "-1" points | 14 | 11
  Change of "0" points | 48 | 59
  Change of "+1" points | 3 | 3
  Change of "+2" points | 0 | 0
  Missing | 0 | 1

47. Secondary Outcome: Change From Baseline to Week 8 in the Disability Assessment Scale for Domain "Hygiene"
Description: as for outcome 40
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 6 | 1
  Change of "-1" points | 16 | 12
  Change of "0" points | 44 | 58
  Change of "+1" points | 3 | 3
  Change of "+2" points | 0 | 0
  Missing | 2 | 1

48. Secondary Outcome: Change From Baseline to Week 12 in the Disability Assessment Scale for Domain "Hygiene"
Description: as for outcome 40
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 4 | 1
  Change of "-1" points | 11 | 12
  Change of "0" points | 50 | 53
  Change of "+1" points | 4 | 7
  Change of "+2" points | 1 | 0
  Missing | 2 | 2

49. Secondary Outcome: Change From Baseline to Final Visit in the Disability Assessment Scale for Domain "Hygiene"
Description: as for outcome 40
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 1
  Change of "-2" points | 2 | 1
  Change of "-1" points | 10 | 9
  Change of "0" points | 50 | 53
  Change of "+1" points | 6 | 9
  Change of "+2" points | 2 | 0
  Missing | 2 | 2

50. Secondary Outcome: Change From Baseline to Week 2 in the Disability Assessment Scale for Domain "Dressing"
Description: as for outcome 40
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 3 | 0
  Change of "-1" points | 16 | 5
  Change of "0" points | 51 | 69
  Change of "+1" points | 2 | 1
  Change of "+2" points | 0 | 0

51. Secondary Outcome: Change From Baseline to Week 4 in the Disability Assessment Scale for Domain "Dressing"
Description: as for outcome 40
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 5 | 2
  Change of "-1" points | 12 | 15
  Change of "0" points | 53 | 54
  Change of "+1" points | 3 | 3
  Change of "+2" points | 0 | 0
  Missing | 0 | 1

52. Secondary Outcome: Change From Baseline to Week 8 in the Disability Assessment Scale for Domain "Dressing"
Description: as for outcome 40
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 3 | 2
  Change of "-1" points | 16 | 13
  Change of "0" points | 48 | 56
  Change of "+1" points | 3 | 3
  Change of "+2" points | 0 | 0
  Missing | 2 | 1

53. Secondary Outcome: Change From Baseline to Week 12 in the Disability Assessment Scale for Domain "Dressing"
Description: as for outcome 40
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 3 | 3
  Change of "-1" points | 16 | 13
  Change of "0" points | 47 | 53
  Change of "+1" points | 4 | 4
  Change of "+2" points | 0 | 0
  Missing | 2 | 2

54. Secondary Outcome: Change From Baseline to Final Visit in the Disability Assessment Scale for Domain "Dressing"
Description: as for outcome 40
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 2 | 2
  Change of "-1" points | 14 | 16
  Change of "0" points | 50 | 51
  Change of "+1" points | 5 | 4
  Change of "+2" points | 0 | 0
  Missing | 2 | 2

55. Secondary Outcome: Change From Baseline to Week 2 in the Disability Assessment Scale for Domain "Limb Position"
Description: as for outcome 40
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 2 | 0
  Change of "-1" points | 22 | 8
  Change of "0" points | 43 | 65
  Change of "+1" points | 5 | 2
  Change of "+2" points | 0 | 0

56. Secondary Outcome: Change From Baseline to Week 4 in the Disability Assessment Scale for Domain "Limb Position"
Description: as for outcome 40
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 7 | 1
  Change of "-1" points | 25 | 10
  Change of "0" points | 37 | 59
  Change of "+1" points | 4 | 4
  Change of "+2" points | 0 | 0
  Missing | 0 | 1

57. Secondary Outcome: Change From Baseline to Week 8 in the Disability Assessment Scale for Domain "Limb Position"
Description: as for outcome 40
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 4 | 1
  Change of "-1" points | 26 | 10
  Change of "0" points | 37 | 61
  Change of "+1" points | 4 | 2
  Change of "+2" points | 0 | 0
  Missing | 2 | 1

58. Secondary Outcome: Change From Baseline to Week 12 in the Disability Assessment Scale for Domain "Limb Position"
Description: as for outcome 40
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 3 | 3
  Change of "-1" points | 19 | 9
  Change of "0" points | 45 | 56
  Change of "+1" points | 3 | 5
  Change of "+2" points | 1 | 0
  Missing | 2 | 2

59. Secondary Outcome: Change From Baseline to Final Visit in the Disability Assessment Scale for Domain "Limb Position"
Description: as for outcome 40
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 0 | 0
  Change of "-2" points | 1 | 3
  Change of "-1" points | 22 | 14
  Change of "0" points | 42 | 51
  Change of "+1" points | 5 | 5
  Change of "+2" points | 1 | 0
  Missing | 2 | 2

60. Secondary Outcome: Change From Baseline to Week 2 in the Disability Assessment Scale for Domain "Pain"
Description: as for outcome 40
Time Frame: Baseline, Week 2
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 1 | 0
  Change of "-2" points | 3 | 0
  Change of "-1" points | 12 | 5
  Change of "0" points | 54 | 69
  Change of "+1" points | 3 | 0
  Change of "+2" points | 0 | 1

61. Secondary Outcome: Change From Baseline to Week 4 in the Disability Assessment Scale for Domain "Pain"
Description: as for outcome 40
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 8 | 2
  Change of "-1" points | 11 | 4
  Change of "0" points | 46 | 67
  Change of "+1" points | 6 | 1
  Change of "+2" points | 0 | 0
  Missing | 0 | 1

62. Secondary Outcome: Change From Baseline to Week 8 in the Disability Assessment Scale for Domain "Pain"
Description: as for outcome 40
Time Frame: Baseline, Week 8
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 4 | 1
  Change of "-1" points | 11 | 7
  Change of "0" points | 49 | 65
  Change of "+1" points | 5 | 0
  Change of "+2" points | 0 | 1
  Missing | 2 | 1

63. Secondary Outcome: Change From Baseline to Week 12 in the Disability Assessment Scale for Domain "Pain"
Description: as for outcome 40
Time Frame: Baseline, Week 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 3 | 0
  Change of "-2" points | 3 | 1
  Change of "-1" points | 10 | 9
  Change of "0" points | 52 | 62
  Change of "+1" points | 3 | 0
  Change of "+2" points | 0 | 1
  Missing | 2 | 2

64. Secondary Outcome: Change From Baseline to Final Visit in the Disability Assessment Scale for Domain "Pain"
Description: as for outcome 40
Time Frame: as for outcome 12
Population: Intention to treat (ITT) as defined as all randomized subjects
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Change of "-3" points | 2 | 0
  Change of "-2" points | 3 | 2
  Change of "-1" points | 11 | 7
  Change of "0" points | 51 | 63
  Change of "+1" points | 4 | 0
  Change of "+2" points | 0 | 1
  Missing | 2 | 2

65. Secondary Outcome: Change From Baseline to Week 4 in the Carer Burden Scale for Domain "Cleaning the Palm of the Affected Hand"
Description: The Carer Burden Scale evaluates the impact of antispastic medication on the physical burden of the carer. It consists of the following items: A=cleaning the palm of the affected hand; B=cutting the fingernails of the affected hand; C=Cleaning the armpit of the affected arm; D=putting the affected arm through the sleeve; E=applying a splint on the affected arm. Each item was assessed on a 5-point Likert scale which values ranges from 0 (=no difficulty) to 4 (=cannot do the task).
Time Frame: Baseline, Week 4
Population: Intention to treat (ITT) as defined as all randomized subjects; missing values were imputed by baseline value, i.e. zero change
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 20
  No longer necessary | 3 | 0
  Less difficult | 15 | 9
  Unchanged | 24 | 38
  More difficult | 5 | 4
  Required for the first time | 0 | 3
  Missing | 0 | 1

66. Secondary Outcome: Change From Baseline to Week 12 in the Carer Burden Scale for Domain "Cleaning the Palm of the Affected Hand"
Description: as for outcome 65
Time Frame: Baseline, Week 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 22
  No longer necessary | 2 | 1
  Less difficult | 12 | 4
  Unchanged | 26 | 38
  More difficult | 7 | 5
  Required for the first time | 0 | 3
  Missing | 0 | 2

67. Secondary Outcome: Change From Baseline to Final Visit in the Carer Burden Scale for Domain "Cleaning the Palm of the Affected Hand"
Description: as for outcome 65
Time Frame: as for outcome 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 27 | 22
  No longer necessary | 2 | 0
  Less difficult | 8 | 4
  Unchanged | 26 | 36
  More difficult | 9 | 5
  Required for the first time | 1 | 6
  Missing | 0 | 2

68. Secondary Outcome: Change From Baseline to Week 4 in the Carer Burden Scale for Domain "Cutting the Fingernails of the Affected Hand"
Description: as for outcome 65
Time Frame: Baseline, Week 4
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 20
  No longer necessary | 0 | 0
  Less difficult | 17 | 12
  Unchanged | 19 | 36
  More difficult | 11 | 5
  Required for the first time | 0 | 1
  Missing | 0 | 1

69. Secondary Outcome: Change From Baseline to Week 12 in the Carer Burden Scale for Domain "Cutting the Fingernails of the Affected Hand"
Description: as for outcome 65
Time Frame: Baseline, Week 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 22
  No longer necessary | 1 | 0
  Less difficult | 12 | 15
  Unchanged | 21 | 26
  More difficult | 13 | 9
  Required for the first time | 0 | 1
  Missing | 0 | 2

70. Secondary Outcome: Change From Baseline to Final Visit in the Carer Burden Scale for Domain "Cutting the Fingernails of the Affected Hand"
Description: as for outcome 65
Time Frame: as for outcome 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 27 | 22
  No longer necessary | 1 | 1
  Less difficult | 12 | 12
  Unchanged | 21 | 26
  More difficult | 12 | 10
  Required for the first time | 0 | 2
  Missing | 0 | 2

71. Secondary Outcome: Change From Baseline to Week 4 in the Carer Burden Scale for Domain "Cleaning the Armpit of the Affected Arm"
Description: as for outcome 65
Time Frame: Baseline, Week 4
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 20
  No longer necessary | 3 | 0
  Less difficult | 11 | 8
  Unchanged | 27 | 38
  More difficult | 4 | 6
  Required for the first time | 2 | 2
  Missing | 0 | 1

72. Secondary Outcome: Change From Baseline to Week 12 in the Carer Burden Scale for Domain "Cleaning the Armpit of the Affected Arm"
Description: as for outcome 65
Time Frame: Baseline, Week 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 22
  No longer necessary | 1 | 2
  Less difficult | 12 | 7
  Unchanged | 25 | 33
  More difficult | 6 | 8
  Required for the first time | 3 | 1
  Missing | 0 | 2

73. Secondary Outcome: Change From Baseline to Final Visit in the Carer Burden Scale for Domain "Cleaning the Armpit of the Affected Arm"
Description: as for outcome 65
Time Frame: as for outcome 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 27 | 22
  No longer necessary | 1 | 2
  Less difficult | 12 | 6
  Unchanged | 23 | 32
  More difficult | 6 | 9
  Required for the first time | 4 | 2
  Missing | 0 | 2

74. Secondary Outcome: Change From Baseline to Week 4 in the Carer Burden Scale for Domain "Putting the Affected Arm Through the Sleeve (e.g., Coat, Shirt, Jacket)"
Description: as for outcome 65
Time Frame: Baseline, Week 4
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 20
  No longer necessary | 2 | 1
  Less difficult | 18 | 11
  Unchanged | 25 | 36
  More difficult | 2 | 4
  Required for the first time | 0 | 2
  Missing | 0 | 1

75. Secondary Outcome: Change From Baseline to Week 12 in the Carer Burden Scale for Domain "Putting the Affected Arm Through the Sleeve (e.g., Coat, Shirt, Jacket)"
Description: as for outcome 65
Time Frame: Baseline, Week 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 22
  No longer necessary | 2 | 3
  Less difficult | 17 | 13
  Unchanged | 24 | 28
  More difficult | 4 | 6
  Required for the first time | 0 | 1
  Missing | 0 | 2

76. Secondary Outcome: Change From Baseline to Final Visit in the Carer Burden Scale for Domain "Putting the Affected Arm Through the Sleeve (e.g., Coat, Shirt, Jacket)"
Description: as for outcome 65
Time Frame: as for outcome 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 27 | 22
  No longer necessary | 3 | 4
  Less difficult | 16 | 10
  Unchanged | 24 | 29
  More difficult | 3 | 6
  Required for the first time | 0 | 2
  Missing | 0 | 2

77. Secondary Outcome: Change From Baseline to Week 4 in the Carer Burden Scale for Domain "Applying a Splint on the Affected Arm"
Description: as for outcome 65
Time Frame: Baseline, Week 4
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 20
  No longer necessary | 1 | 1
  Less difficult | 5 | 1
  Unchanged | 40 | 51
  More difficult | 1 | 0
  Required for the first time | 0 | 1
  Missing | 0 | 1

78. Secondary Outcome: Change From Baseline to Week 12 in the Carer Burden Scale for Domain "Applying a Splint on the Affected Arm"
Description: as for outcome 65
Time Frame: Baseline, Week 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 26 | 22
  No longer necessary | 2 | 1
  Less difficult | 2 | 2
  Unchanged | 42 | 46
  More difficult | 1 | 0
  Required for the first time | 0 | 2
  Missing | 0 | 2

79. Secondary Outcome: Change From Baseline to Final Visit in the Carer Burden Scale for Domain "Applying a Splint on the Affected Arm"
Description: as for outcome 65
Time Frame: as for outcome 12
Population: as for outcome 65
Measure: Number; unit: Participants
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No carer | 27 | 22
  No longer necessary | 3 | 1
  Less difficult | 1 | 2
  Unchanged | 41 | 45
  More difficult | 1 | 1
  Required for the first time | 0 | 2
  Missing | 0 | 2

ADVERSE EVENTS:
Time Frame: All SAEs/AEs during Double-Blind Period After Injection.
Description: The table of "Other Adverse Events" includes all AEs, both non serious and serious. Only results and AEs of the Double-Blind Period are given as the Open-Label Extension Period was a non-controlled study. The investigator asked the patient for AEs systematically at each visit.
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/73 | 1/75
Other Adverse Events (participants affected / at risk) | 10/73 | 5/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (N=73) | Placebo (N=75)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (N=73) | Placebo (N=75)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 wks before submission. Sponsor to give written opinion within 30 d. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.